CLINICAL TRIAL: NCT06085092
Title: Evaluating Open Weighing and Blind Weighing in the Treatment of Adolescents and Young Adults With Eating Disorders
Brief Title: Open vs. Blind Weighing Study In Adolescents and Young Adult With Eating Disorders
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Jamal Essayli, Assistant Professor of Pediatrics and Psychiatry & Behavioral Health, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22718
Record Dates: First submitted 2023-10-05; First posted 2023-10-16 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Eating Disorders; Anorexia Nervosa
Keywords: Eating Disorders; Anorexia Nervosa
MeSH Terms: conditions — Feeding and Eating Disorders; Anorexia Nervosa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Open weighing (Experimental): The open-weighing intervention aims to challenge beliefs about weight gain. The study coordinator (SC) will explain open weighing, discuss any concerns you have about your weight, and construct a weight graph with the number of weeks on the x-axis and weight in pounds on the y-axis. The SC will help identify beliefs about gaining weight, which will be written on a Feared Outcomes Form. The SC will ask you to predict your weight, mark the weight prediction on the graph, weigh you on a standing scale, record your weight, and discuss your responses to seeing your weight, including any reasons for a difference between your predicted and actual weight. Each week, the SC will graph your actual and predicted weights over time and discuss anything that you are learning from this process. The SC will ask you to complete the Feared Outcomes Form once per day over the next week, review it each week, and talk to you about what you are learning from this process.
  Interventions: Behavioral: Open weighing
- Blind weighing (Active Comparator): The blind weighing intervention aims to help you see self-weighing as an eating disorder symptom that you should stop, and that weight is not important to your identity or selfesteem. To do this, the study coordinator will explain why blind weighing might be helpful. You will then be asked to step backwards on a standing scale. The study coordinator will record your weight, but will not share your weight information with you. The study coordinator will discourage you from thinking or talking about your weight.
  Interventions: Behavioral: Blind weighing

INTERVENTIONS:
Behavioral: Open weighing — The open-weighing intervention aims to challenge beliefs about weight gain. The study coordinator (SC) will explain open weighing, discuss any concerns you have about your weight, and construct a weight graph with the number of weeks on the x-axis and weight in pounds on the y-axis. The SC will help identify beliefs about gaining weight, which will be written on a Feared Outcomes Form. The SC will ask you to predict your weight, mark the weight prediction on the graph, weigh you on a standing scale, record your weight, and discuss your responses to seeing your weight, including any reasons for a difference between your predicted and actual weight. Each week, the SC will graph your actual and predicted weights over time and discuss anything that you are learning from this process. The SC will ask you to complete the Feared Outcomes Form once per day over the next week, review it each week, and talk to you about what you are learning from this process.
  Arms: Open weighing
Behavioral: Blind weighing — The blind weighing intervention aims to help you see self-weighing as an eating disorder symptom that you should stop, and that weight is not important to your identity or self-esteem. To do this, the study coordinator will explain why blind weighing might be helpful. You will then be asked to step backwards on a standing scale. The study coordinator will record your weight but will not share your weight information with you. The study coordinator will discourage you from thinking or talking about your weight.
  Arms: Blind weighing

SUMMARY:
Current treatments for adolescents and young adults (AYAs) with eating disorders (EDs) do not effectively address a central ED symptom - anxiety about weight gain - which contributes to poor outcomes. The proposed study evaluates the feasibility, acceptability, efficacy, and underlying mechanisms of an enhanced version of "open weighing," a cognitive-behavioral intervention designed to target anxiety about weight gain in AYAs with EDs. Understanding how to better treat AYAs with EDs, and identifying the mechanisms by which interventions lead to improvement, will aid in the development of more effective and personalized treatments, ultimately improving the lives of AYAs with EDs.

DETAILED DESCRIPTION:
The proposed study evaluates the feasibility, acceptability, efficacy, and underlying mechanisms of an enhanced version of "open weighing" (OW), a cognitive-behavioral intervention designed to target anxiety about weight gain in adolescents and young adults (AYAs) with eating disorders (EDs). OW will be compared to an alternative intervention, "blind weighing" (BW), in which individuals are discouraged from seeing, thinking, or talking about their weight. Understanding how to better treat AYAs with EDs, and identifying the mechanisms by which interventions lead to improvement, will aid in the development of more effective and personalized treatments, ultimately improving the lives of AYAs with EDs.

Aim 1. Evaluate the feasibility and acceptability of OW and BW for AYAs with EDs.

Hypothesis 1.1: Both OW and BW will be feasible, with no significant differences in rates of recruitment or retention.

Hypothesis 1.2: Both treatments will be rated as highly acceptable, with no significant differences in measures evaluating the acceptability or attitudes about OW and BW.

Aim 2. Test the efficacy of OW and BW. Hypothesis 2.1: OW will result in significantly greater improvements in body mass index and ED symptomatology than BW.

Hypothesis 2.2: OW will result in significantly greater decreases in anxiety about weight gain than BW.

Aim 3. Identify anxiety about weight gain as a key mechanism to target in the treatment of AYAs with EDs.

Hypothesis 3.1: Across both conditions, greater reductions in anxiety about weight gain will be associated with better outcomes at discharge.

ELIGIBILITY:
Inclusion Criteria:

* Participants must be English speakers.
* Participants must be between the ages of 12 - 24 years who have been admitted to either the adolescent or young adult Partial Hospital Program (PHP) for eating disorders (EDs) at Penn State Hershey.
* Participants must also present with an eating disorder (ED) diagnosis that is characterized by anxiety about weight gain, such as anorexia nervosa (AN), Bulimia nervosa (BN), or their subthreshold presentations captured under the other specific feeding or eating disorder (OSFED) category.

Exclusion Criteria:

* Participants will be excluded if they are above the age of 24 or below the age of 12 years.
* Participants who have been identified as non-English speakers.
* Participants with cognitive impairment will also be excluded from participation.
* Potential participants will be excluded if they do not meet the diagnostic inclusion criteria noted above.
* individuals with a diagnosis of avoidant/restrictive food intake disorder, as these individuals do not experience anxiety about weight gain will be excluded.

Ages: 12 Years to 24 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 70 (Estimated)
Dates: Start 2023-10-31 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Eating Disorder Examination - Self-Report Questionnaire (EDE-Q) | Admission-Baseline
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire. It was designed to assess the range, frequency, and severity of behaviors associated with a diagnosis of an eating disorder. A total score is obtained by summing the four subscales scores and dividing the total by the number of subscales. The score of items are calculated and range from 0 to 36. The higher score indicate greater ED symptoms.
Fear of Food Measure (FOFM) | Admission Baseline
  The Fear of Food Measure (FORM) is a 23-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. Each item is scored on a 1-7 scale. The questionnaire range from 23 to 161 meaning 23: no fear of food and 161 meaning severe fear of food.
Body Shape Questionnaire (BSQ) | Admission- Baseline
  The BSQ is a self-reported measurement of the body shape concerns typical of bulimia nervosa and anorexia nervosa. The questionnaire has 34 items scored from 0 to 6 points (least and most impaired, respectively), with the sum of the questions giving a range from 0 to 204.
Clinical Impairment Assessment (CIA) | Admission- Baseline
  The Clinical Impairment Assessment Questionnaire (CIA) is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features and focuses on the past 28 days. The 16 items cover impairment in domains of life that are typically affected by eating disorder psychopathology: mood and self-perception, cognitive functioning, interpersonal functioning, and work performance. The response are scored 0,1,2 and 3 with a higher rating indicating a higher level of impairment. The total range is between 0 and 48.
Eating Disorder Fear Questionnaire (EDFQ) | Admission_Baseline
  The Eating Disorder Fear Questionnaire (EDFQ) is a 20-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. The response range between 1 to 7 with a total range of 20 to 140. The higher rating indicating a higher severe impairment.
Eating Disorder-15 (ED 15) | Admission_Baseline
  The Eating Disorder-15 (ED-15) is a 15-item measure designed to assess eating psychopathology levels over the preceding week. The 10 items scored from 0 to 6 points (least and most impaired, respectively), with the sum of the questions giving a range from 0 to 6. The additional 5 items focused on the number of days individuals participated in a given behavior, such as the use of laxatives and restrictive eating.
Body Image States Scale (BISS) | Admission_Baseline
  The Body Image State Scale (BISS) is a 6-item measure designed to assess body dissatisfaction. The questionnaire is rated on a seven-point scale ranging from "very satisfied" to very dissatisfied".
Approach / Avoidance of weighing Questionnaire (AAWQ) | Admission_Baseline
  The Approach / Avoidance of Weighing Questionnaire (AAWQ) is a 9-item measure designed to assess approach and avoidance weighing tendency. The three descriptive items are not included in the approach/avoidance weighing tendencies calculation. Items 1-3 correspond to approach weighing tendency, and items 4-6 correspond to avoidance weighing tendency. Items are scored as follows for both subscales: Totally true of me = 5; Somewhat true of me = 4; Neither true nor untrue of me = 3; Somewhat untrue of me = 2; Totally untrue of me = 1. Items 1-3 are summed to provide the approach weighing tendency subscale and items 4-6 are summed to provide the avoidance weighing tendency subscale, with scores ranging from 3-15. Higher scores on each subscale indicate a higher degree of that subscale's weighing tendency.
Eating Disorder Examination - Self-Report Questionnaire (EDE-Q) | Discharge: No longer than 60 weeks
  The Eating Disorder Examination Questionnaire (EDE-Q) is a 28-item self-report questionnaire. It was designed to assess the range, frequency, and severity of behaviors associated with a diagnosis of an eating disorder. A total score is obtained by summing the four subscales scores and dividing the total by the number of subscales. The score of items are calculated and range from 0 to 36. The higher score indicate greater ED symptoms.
Fear of Food Measure (FOFM) | Discharge: No longer than 60 weeks
  The Fear of Food Measure (FORM) is a 23-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. Each item is scored on a 1-7 scale. The questionnaire range from 23 to 161 meaning 23: no fear of food and 161 meaning severe fear of food.
Body Shape Questionnaire (BSQ) | Discharge: No longer than 60 weeks
  The BSQ is a self-reported measurement of the body shape concerns typical of bulimia nervosa and anorexia nervosa. The questionnaire has 34 items scored from 0 to 6 points (least and most impaired, respectively), with the sum of the questions giving a range from 0 to 204.
Clinical Impairment Assessment (CIA) | Discharge: No longer than 60 weeks
  The Clinical Impairment Assessment Questionnaire (CIA) is a 16-item self-report measure of the severity of psychosocial impairment due to eating disorder features and focuses on the past 28 days. The 16 items cover impairment in domains of life that are typically affected by eating disorder psychopathology: mood and self-perception, cognitive functioning, interpersonal functioning, and work performance. The response are scored 0,1,2 and 3 with a higher rating indicating a higher level of impairment. The total range is between 0 and 48.
Eating Disorder Fear Questionnaire (EDFQ) | Discharge: No longer than 60 weeks
  The Eating Disorder Fear Questionnaire (EDFQ) is a 20-item self-report questionnaire. It examines the participant's severity of behaviors associated with a diagnosis of an eating disorder. The response range between 1 to 7 with a total range of 20 to 140. The higher rating indicating a higher severe impairment.
Eating Disorder-15 (ED-15) | Discharge: No longer than 60 weeks
  The Eating Disorder-15 (ED-15) is a 15-item measure designed to assess eating psychopathology levels over the preceding week. The 10 items scored from 0 to 6 points (least and most impaired, respectively), with the sum of the questions giving a range from 0 to 6. The additional 5 items focused on the number of days individuals participated in a given behavior, such as the use of laxatives and restrictive eating.
Body Image State Scale (BISS) | Discharge: No longer than 60 weeks
  The Body Image State Scale (BISS) is a 6-item measure designed to assess body dissatisfaction. The questionnaire is rated on a seven-point scale ranging from "very satisfied" to very dissatisfied".
Approach / Avoidance of Weighing Questionnaire (AAWQ) | Discharge: No longer than 60 weeks
  The Approach / Avoidance of Weighing Questionnaire (AAWQ) is a 9-item measure designed to assess approach and avoidance weighing tendency. The three descriptive items are not included in the calculation of approach/avoidance weighing tendencies. The items 1-3 correspond to approach weighing tendency, and items 4-6 correspond to avoidance weighing tendency. Items are scored as follows for both subscales: Totally true of me = 5; Somewhat true of me = 4; Neither true nor untrue of me = 3; Somewhat untrue of me = 2; Totally untrue of me = 1. Items 1-3 are summed to provide the approach weighing tendency subscale and items 4-6 are summed to provide the avoidance weighing tendency subscale, with scores ranging from 3-15. Higher scores on each subscale indicate a higher degree of that subscale's weighing tendency.

SECONDARY OUTCOMES:
Personal Reactions to the Rationale questionnaire (PRR) | Admission-Baseline
  The Personal Reactions to the Rationale questionnaire (PRR) is a 16-item that assesses participants' attitudes about Open weighing (OW) and Blind weighing (BW). The response range between 1 to 7 with a total range of 24 to 168. The higher rating indicate participants' attitudes about OW and BW.
Credibility Scale (CS) | Admission-Baseline
  Credibility Scale (SC) is a 8-item that assesses participants' attitudes about Open weighing (OW) and Blind weighing (BW). The response range between 1 to 7 with a total range of 24 to 168. The higher rating indicate participants' attitudes about OW and BW.

CONTACTS AND LOCATIONS:
Overall Officials: Jamal Essayli, Ph.D, Principal Investigator — Penn State University
Locations (1):
- 905 W Govener Rd, Hershey, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No